CLINICAL TRIAL: NCT05316363
Title: Efficacy and Safety of Osteopathic Manipulative Treatment on Asthmatics
Brief Title: Efficacy and Safety of OMT on Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jesus Sanchez, Assistant Dean of Academic Affairs, Professor of NMM/OMM & Family Medicine, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/IRB/090
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Asthma
Keywords: OMT
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Randomized into two groups: Standard asthmatic care with OMT intervention and standard asthmatic care with no OMT.
Who Masked: Care Provider, Investigator
Masking Description: Care providers were not involved in any data analysis and the investigator was also blind to the assignment and outcomes assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT Intervention Arm (Experimental): Patients treated with 4 techniques for 8 minutes in the supine position. OMT systematically administered to address the 4 body regions - cervical spine, thoracic spine, ribs and diaphragm. The techniques utilized for this study include: suboccipital release, diaphragmatic release, rib raising and paraspinal inhibition of the thoracic spine. Each technique administered for approximately 2 minutes.
  Interventions: Other: OMT
- Control (No Intervention): Patients lie supine on the treatment table and rested quietly for a total of 8 minutes.

INTERVENTIONS:
Other: OMT — Suboccipital Release - Finger pads are placed onto suboccipital musculature and a smooth, gentle, and rhythmic laterocephalad traction is applied to reduce muscle tension.
  Paraspinal Inhibition - Hands are placed under the patient's thoracolumbar spine and contract the erector spinae tissue to draw the thoracolumbar spine into extension and hold until relaxation is felt.
  Rib Raising - Hands are placed under the subject's thorax and contact the rib angles with finger pads. Fingers are flexed while adding an anteriolateral traction directed at the rib angle while maintaining neutral wrists. Arms are used as a lever by leaning forward thus creating a fulcrum with the treatment table with a smooth, rhythmic motion. This motion is repeated several times throughout the entire thoracic region, unilaterally and then switch sides.
  Diaphragm Release - Hands apply a gentle pressure until a barrier or point of ease of the fascia is felt and hold that position until tissue response is felt.
  Arms: OMT Intervention Arm

SUMMARY:
This is a pilot study in which the objective is to determine the feasibility of a randomized clinical trial investigating the safety and efficacy of OMT as an adjunctive treatment for patients with mild to moderate asthma compared to the same patient population without the use of OMT. OMT may be able to correct anatomical dysfunctions that contribute to increased symptoms in asthmatic patients. OMT's effect on asthma will be demonstrated by symptomatology reporting, frequency of medication use, and pulmonary function tests.

DETAILED DESCRIPTION:
Asthma is a leading cause of activity limitation and healthcare burden in the United States of America. The asthmatic population is in need of treatments that target reducing asthma symptoms, reduce the need for medication, and improve lung functionality. As of today, there are not many studies investigating the efficacy and safety of osteopathic manipulative treatment (OMT) on asthmatic patients. This is a pilot study in which the objective is to determine the feasibility of a randomized clinical trial investigating the safety and efficacy of OMT as an adjunctive treatment for patients with mild to moderate asthma compared to the same patient population without the use of OMT. Subjects will be randomized into either a control group or an intervention group where OMT will be used in conjunction with standard asthmatic treatment. Subjective and objective measurements will be taken including the Asthma Control Test (ACT) questionnaire, peak flow, spirometry, pulse oximetry, and chest/diaphragmatic excursion measurements. Measurements will be compared from baseline, before the first treatment and at the follow-up visit after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with mild to moderate asthma (Episodic symptoms included were airflow obstruction or airway hyper-responsiveness, and airflow obstruction that was at least partially reversible (based upon an increase in FEV1 or greater than or equal to 12% from baseline or by an increase of at least 10% of predicted FEV1 after inhalation of a short-acting bronchodilator)

Exclusion Criteria:

* pneumonia
* COPD as a primary diagnosis
* pulmonary fibrosis
* smoking history
* inability to perform pulmonary function tests
* history of recent myocardial infarction or heart disease
* unable to respond to the questionnaire
* unable to provide informed consent
* pregnant
* using muscle relaxants
* Any contraindications to OMT such as: known bone metastases, severe osteoporosis, osteomyelitis, or fracture

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) Score | Between baseline and 5 weeks
  Determine the efficacy of adjunctive OMT treatment when compared to standard care in the reduction of symptomatology of dyspnea, wheezing and bronchoconstriction and decrease medication use as measured by the Expert Panel Report 3 and Global Initiative for Asthma Monitoring Asthma Control Test (ACT) questionnaire which is scored on a range from 5 to 25 with higher scores indicating better control of asthma symptoms.

SECONDARY OUTCOMES:
Morphological Measurements of Chest and Diaphragm Excursion | Between baseline and 5 weeks
  Chest wall and diaphragm excursion measurements were obtained to assess wall and diaphragm motion during respiration at three different levels: The anterior landmarks were the third intercostal space, xiphoid process and superior aspect of umbilicus which corresponded with the posterior landmarks of the transverse processes of T5, T10 and T12 vertebrae, respectively for participants with and without OMT.
Pulse Oximetry (Pulse Rate) | Between baseline and 5 weeks
  Pulse rate in beats per minute (BPM) was compared between subjects who received OMT as compared to subjects who only received standard care.
Pulse Oximetry (Blood O2 Saturation Levels) | Between baseline and 5 weeks
  Blood O2 Saturation levels as measured by a pulse oximeter as a percentage was compared between subjects that received OMT versus those treated with only standard care.
Spirometry Readings: Forced Expiratory Volume in One Second (FEV1) | Between baseline and 5 weeks
  Forced expiratory volume in one second was reported as volume of air expired in one second in subjects who received OMT as compared to subjects who only received standard care.

IPD SHARING:
Plan to Share IPD: No